CLINICAL TRIAL: NCT00422331
Title: Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter, Efficacy and Safety Study of Lithium in Bipolar I Disorder
Brief Title: Safety and Efficacy Study of Lithium in Bipolar Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JDS Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDS04004; Lithium TEAM-1 Study
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Bipolar Disorder; Mania
Keywords: Bipolar I Disorder; Bipolar Disorder; Lithium
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Lithium Carbonate

INTERVENTIONS:
Drug: Lithium Carbonate Capsule

SUMMARY:
The purpose of this study is to determine whether Lithium is safe and effective in the treatment of Bipolar I Disorder subjects with symptoms of acute mania.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar 1 Disorder;
* Hospitalized or in the process of being hospitalized for a manic or mixed episode

Exclusion Criteria:

* History of rapid cycling;
* History of hypersensitivity or adverse reaction to lithium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in YMRS score

SECONDARY OUTCOMES:
change from baseline in CGI-BP score
change from baseline in MADRS score

CONTACTS AND LOCATIONS:
Locations (1):
- JDS Pharmaceuticals, New York, New York, United States